CLINICAL TRIAL: NCT00981071
Title: The Time of Positive Conversion of Interferon-γ Releasing Assay After Tuberculosis Exposure
Status: Completed | Type: Observational
Sponsor: Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Sei Won Lee/Division chief of pulmonology, Armed Forces Capital Hospital
Other Study IDs: QFTconversion
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; QuantiFERON; Outbreak; Conversion
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A platoon with TB outbreak

SUMMARY:
The aim is to evaluate the time of positive conversion after exposure to smear positive pulmonary tuberculosis (TB) in a platoon of Korean military, a closed communal setting.

DETAILED DESCRIPTION:
In a platoon where TB outbreak occurred, we performed low dose chest CT (LDCT), QuantiFERON-TB gold in tube (QFT) and two-step (0, 4weeks) TST for outbreak investigation. We perform QFT at 0, 2, 4, 8 and 12 weeks after initial investigation for soldiers with negative QFT results, and soldiers with positive QFT and normal LDCT took isoniazid and rifampin for 3 months as treatment of latent TB.

ELIGIBILITY:
Inclusion Criteria:

* All soldiers who assigned to the military platoon where a tuberculosis outbreak occurred

Exclusion Criteria:

* Soldiers who could not complete study or refused the study protocol

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A military unit in South Korean Army
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital